CLINICAL TRIAL: NCT04397432
Title: Synergistic Real-world Study and Evidence-based Medicine Evaluation of Elemene Combined With Tyrosine Kinase Inhibitors（TKIs）in the Treatment of Advanced Non-small Cell Lung Cancer（NSCLC）：Retrospective Study
Brief Title: Synergistic Effect of Elemene Plus TKIs Compared With TKIs in EGFR-mutated Advanced NSCLC：Retrospective Study
Acronym: SELECT-1
Status: Active, not recruiting | Type: Observational
Sponsor: Tian Xie (Other)
Collaborators: LinkDoc Technology (Beijing) Co. Ltd. (Industry)
Responsible Party: Sponsor-Investigator, Tian Xie, Professor, Hangzhou Normal University
Organization: Hangzhou Normal University (Other)
Other Study IDs: HangzhouNU
Record Dates: First submitted 2020-05-18; First posted 2020-05-21 (Actual); Last update posted 2023-12-27 (Actual); Status verified 2023-12

CONDITIONS: Carcinoma, Non-Small-Cell Lung
Keywords: Elemene, TKI, EGFR, Real world study
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Elemene plus TKIs: This is a real-world study, we just record the patient's medication who used Elemene Injectable Emulsion and/or Elemene Oral Emulsion plus TKIs. First, second or third generation TKIs were all available, such as Erlotinib, Gefitinib, Icotinib, Afatinib, Dacomitinib, and Osimertinib.
- TKIs only: This is a real-world study, we just record the patient's medication who used TKIs only. First, second or third generation TKIs were all available, such as Erlotinib, Gefitinib, Icotinib, Afatinib, Dacomitinib, and Osimertinib.

SUMMARY:
This is a nationwide, multicenter and retrospective cohort study. The purpose of this study is to evaluate the synergistic effect and safety of Elemene plus TKIs in EGFR-mutated advanced non-small cell lung cancer.

DETAILED DESCRIPTION:
About 9.2%-45.8% of Chinese patients with Non-small cell lung cancer were positive for EGFR gene mutation. Gefitinib, Erlotinib, Icotinib, Afatinib showed efficacy superior to that of chemotherapy in the treatment of EGFR mutation positive advanced NSCLC, and lower rates of serious adverse events. However, after a median of 8 to 13 months of disease control, patients ultimately progress due to acquired resistance of EGFR-TKIs. Elemene, a chemotherapeutic isolated from the Chinese medicinal herb Rhizoma Zedoariae, has been shown to have a comprehensive anti-tumor effect and the potential effect on reversing drug resistance.

The study is a real-world study and the case records of patients with advanced non-small cell lung cancer who visited the research centers from January 2014 to December 2017 and met the inclusion criteria will be collected. Medical data including patient demographic, tumor characteristics, laboratory examination, history of treatments, adverse reactions, and so on will be extracted to evaluate the synergistic effect and safety of Elemene plus TKIs in EGFR-mutated advanced non-small cell lung cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed advanced non-small cell lung cancer(stage IIIB~IV).
2. Patients with EGFR mutation.
3. Received EGFR-TKIs at least once.
4. Received Elemene Injectable Emulsion and/or Elemene Oral Emulsion at least once ( only for Elemene plus TKIs group).
5. Completeness of important outcome measures and medical records related to the study.

Exclusion Criteria:

1. Accompanied by other active tumors.
2. The researchers did not consider it appropriate to participate in this study for other reasons.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with advanced non-small cell lung cancer and EGFR mutation who visited the research centers from January 2014 to December 2017 and received TKIs therapy with or without Elemene.
Sampling Method: Non-Probability Sample
Enrollment: 878 (Actual)
Dates: Start 2020-08-28 (Actual); Primary Completion 2023-04-30 (Actual); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
OS | June 2021
  OS was defined as the interval from the date of the administration of the first-dose TKIs to date of death from any cause, or the date of last known follow-up alive.

SECONDARY OUTCOMES:
PFS | June 2021
  PFS was defined as the interval from date of the administration of the first-dose TKIs to the date of first evidence of disease progression or death, whichever occurs first. Disease progression was defined according to RECIST 1.1.
ORR | June 2021
  ORR was defined as the percentage of participants with best overall response (BOR) of complete response (CR) or partial response (PR) based on RECIST 1.1.
DCR | June 2021
  Disease Control Rate (DCR) = Complete Response (CR) + Partial Response (PR) + Stable Disease (SD) as defined by RECIST 1.1.
KPS score | June 2021
  Performance status were measured by Karnofsky Performance Scale (KPS).
ECOG score | June 2021
  Eastern Cooperative Oncology Group (ECOG) performance status adopted the zubrod-ecog-who scoring standard.
Incidence and severity of AE or SAE | Start of treatment until 30 days after the last dose.
  Any untoward medical occurrence in a patient or clinical investigation subject administered a pharmaceutical product and which does not necessarily have to have a causal relationship with this treatment.
  A serious adverse event (experience) or reaction is any untoward medical occurrence that at any dose: results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, or is a congenital anomaly/birth defect.

CONTACTS AND LOCATIONS:
Overall Officials: Ziping Wang, PhD, Principal Investigator — Peking University Cancer Hospital & Institute
Locations (19):
- China (19):
  - Affiliated Hospital of Nantong University, Nantong, Jiangsu
  - Panjin Central Hospital, Panjin, Liaoning
  - Shenyang Tenth People's Hospital, Shenyang, Liaoning
  - The Second People's Hospital of Yangcheng County, Jincheng, Shanxi
  - Sichuan Academy of Medical Sciences · Sichuan Provincial People's Hospital, Chengdu, Sichuan
  - Hangzhou Cancer Hospital, Hangzhou, Zhejiang
  - Tongde Hospital of Zhejiang Province, Hangzhou, Zhejiang
  - Zhejiang Hospital, Hangzhou, Zhejiang
  - Zhejiang Xiaoshan Hospital, Hangzhou, Zhejiang
  - Hangzhouwan Hospital, Ningbo, Zhejiang
  - Dongfang Hospital Beijing University of Chinese Medicine, Beijing
  - Beijing Cancer Hospital, Beijing
  - Cancer Hospital Chinese Academy of Medical Sciences, Beijing
  - Cancer Hospital of Huanxing Chaoyang District Beijing, Beijing
  - Chongqing University Cancer Hospital, Chongqing
  - Longhua Hospital Affiliated to Shanghai University of Traditional Chinese Medicine, Shanghai
  - Shuguang Hospital Affiliated to Shanghai University of Traditional Chinese Medicine, Shanghai
  - Tianjin Academy of Traditional Chinese Medicine Affiliated Hospital, Tianjin
  - Tianjin Medical University General Hospital, Tianjin

IPD SHARING:
Plan to Share IPD: Undecided